CLINICAL TRIAL: NCT06284954
Title: A Phase 2, Randomized, Double-Blinded, Placebo-Controlled, Multicenter Study to Evaluate the Safety, Tolerability, and Efficacy of Empasiprubart in Adults With Dermatomyositis
Brief Title: A Study to Evaluate Safety and Efficacy of Empasiprubart in Adults With Dermatomyositis
Acronym: empacific
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARGX-117-2301; 2023-508337-14 (Other: CTIS number)
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Dermatomyositis; Myositis
MeSH Terms: conditions — Dermatomyositis; Myositis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Empasiprubart (Experimental): Patients receiving Empasiprubart IV
  Interventions: Biological: Empasiprubart IV
- Placebo (Placebo Comparator): Patients receiving Placebo IV
  Interventions: Other: Placebo IV

INTERVENTIONS:
Biological: Empasiprubart IV — Intravenous infusion with Empasiprubart IV
  Other Names: ARGX-117
  Arms: Empasiprubart
Other: Placebo IV — Intravenous infusion with Placebo IV
  Arms: Placebo

SUMMARY:
This study will evaluate the safety and efficacy of empasiprubart compared with placebo in adult participants with dermatomyositis (DM).

The study duration will be approximately 92 weeks for all participants. After the screening period, eligible participants will be randomized in a 2:1 ratio to receive either empasiprubart or placebo, respectively, during the treatment period (duration of 25 weeks). At the end of the treatment period, all the participants will enter a safety follow-up period (duration of 65 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years of age and the local legal age of consent for clinical studies when signing the Informed Consent Form
* Is capable of providing signed informed consent and complying with protocol requirements
* Agrees to use contraceptive measures consistent with local regulations and women of child-bearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test before receiving the study drug
* Has a clinical diagnosis of dermatomyositis or juvenile dermatomyositis. The diagnosis date for juvenile dermatomyositis should be ≤5 years before screening
* Has active muscle disease associated with classic dermatomyositis or juvenile dermatomyositis at screening and before the first study drug adminisitration and at least 1 of the following: elevated levels of creatine kinase, aldolase, lactate dehydrogenase, aspartate aminotransaminase or alanine aminotransferase at screening; or electromyography ≤18 weeks before the first study drug administration; or an MRI depicting active muscle inflammation ≤18 weeks before the first study drug administration; or muscle biopsy demonstrating signs of active inflammation ≤18 weeks before the first study drug administration
* Has at least mild skin disease at screening
* Complies with the permitted background dermatomyositis treatment requirements at screening
* Has had immunization with the first meningococcal, pneumococcal, and the single Haemophilus influenza type B vaccine ≥14 days before the first study drug administration

Exclusion Criteria:

* Known autoimmune disease or any medical condition that would interfere with an accurate assessment of clinical symptoms of dermatomyositis or puts the participant at undue risk
* Naïve to standard dermatomyositis treatment according to local recommendations
* History of malignancy unless considered cured by adequate treatment with no evidence of recurrence for ≥3 years before the first study drug administration. Adequately treated participants with the following cancers can be included at any time: Basal cell or squamous cell skin cancer; Carcinoma in situ of the cervix; Carcinoma in situ of the breast; Incidental histological findings of prostate cancer
* Clinically significant active infection that is not sufficiently resolved before the first study drug administration in the investigator's opinion
* Positive serum test at screening for active infection with any of the following: Hepatitis B virus, Hepatitis C virus, HIV
* Clinically significant disease, recent major surgery, or intention to have major surgery during the study; or any other medical condition that, in the investigator's opinion, would confound the results of the study or put the participant at undue risk
* Current participation in another interventional clinical study
* Known hypersensitivity to the study drug or any of its excipients
* History (within 12 months before screening) of or current alcohol, drug, or medication abuse, as assessed by the investigator
* Pregnant or lactating state or intending to become pregnant during the study
* Previous participation in an empasiprubart clinical study with at least 1 dose of study drug received
* Known complement component deficiency as assessed by the investigator
* Change in dermatomyositis physical therapy or exercise program from ≤4 weeks before screening
* Inflammatory or non-inflammatory myopathies other than dermatomyositis, such as drug-induced or endocrine-induced myositis, infective myositis, polymyositis, immune-mediated necrotizing myopathy, inclusion body myositis, overlap myositis, metabolic myopathies, or muscle dystrophies
* Paraneoplastic dermatomyositis secondary to malignancy
* Glucocorticoid-induced myopathy
* Severe muscle damage
* Extensive or severe calcinosis
* Interstitial lung disease with at least 1 of the following: forced vital capacity (FVC) ≤60%; supplemental oxygen therapy; rapidly progressing uncontrolled interstitial lung disease; moderate or severe interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 90 weeks
Percentage of participants discontinuing investigational medicinal product (IMP) due to an adverse event (AE) | Up to 25 weeks

SECONDARY OUTCOMES:
Mean TIS | Up to 25 weeks
  The Total Improvement Score (TIS) assesses minimal, moderate, and major clinical response categorically or continuously using American College of Rheumatology and European League Against Rheumatism (ACR/EULAR) criteria.

CONTACTS AND LOCATIONS:
Locations (28):
- United States (9):
  - Profound Research LLC, Oceanside, California
  - Omega Research Debary, LLC, DeBary, Florida
  - University of Florida Health (UF) - Endocrinology - Medical Specialties - Medical Plaza, Gainesville, Florida
  - Homestead Associates in Research, Inc., Homestead, Florida
  - Life Clinical Trials, Margate, Florida
  - Advance Medical Research Center, Miami, Florida
  - Integral Rheumatology and Immunology Specialists (IRIS), Plantation, Florida
  - D and H Tamarac Research, LLC Center, Tamarac, Florida
  - Wright State Physicians Health Center, Dayton, Ohio
- Georgia (6):
  - V.Tsitlanadze Scientific Practical Reumatology Center, Tbilisi
  - The First University Clinic of Tbilisi State Medical University, Tbilisi
  - Institute of Clinical Cardiology, Ltd, Tbilisi
  - Jerarsi Clinic, Tbilisi
  - Mtskheta street Clinic, Tbilisi
  - The First Medical Center, Tbilisi
- Greece (3):
  - National and Kapodistrian University of Athens (NKUA) - University General Hospital Attikon, Athens
  - Andreas Syggros Hospital of Skin and Venereal Diseases - University Dermatology and Venereology, Athens
  - General Hospital of Thessaloniki Papageorgiou, Thessaloniki
- Italy (2):
  - Azienda Ospedaliera Universitaria Pisana, Pisa
  - Fondazione Policlinico Universitario Campus Bio-Medico, Rome
- Moldova (2):
  - Timofei Mosneaga Republican Clinical Hospital, Chisinau
  - Institute of Cardiology, Chisinau
- Poland (3):
  - Nova Reuma Domyslawska i Rusilowicz- Spolka Partnerska Lekarza Reumatologa i Fizjoterapeuty, Bialystok
  - Prywatna Praktyka Lekarska Prof. UM dr Hab. Med. Pawel Hrycaj, Poznan
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wroclawiu, Wroclaw
- Spain (3):
  - Parc de Salut Mar - Hospital del Mar, Barcelona
  - Hospital Quironsalud Infanta Luisa, Seville
  - Hospital Universitario Rio Hortega, Valladolid

IPD SHARING:
Plan to Share IPD: No